CLINICAL TRIAL: NCT02520102
Title: A Phase II Open Label Study of Sargramostim Among Patients Receiving Myelosuppressive Induction Chemotherapy for Acute Myelogenous Leukemia
Brief Title: Open Label Study of Sargramostim Among Patients Receiving Myelosuppressive Induction Chemotherapy for Acute Myelogenous Leukemia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Company has fulfilled post-marketing requirements
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTS13932; U1111-1148-1183 (Other: UTN)
Record Dates: First submitted 2015-08-07; First posted 2015-08-11 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-03

CONDITIONS: Acute Myeloid Leukemia NOS
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- sargramostim (Experimental): Sargramostim is administered daily until the absolute neutrophil count (ANC) equals or exceeds 1500/mm^3 for 3 consecutive measurements or up to 42 days post-induction chemotherapy.
  Interventions: Drug: sargramostim GZ402664

INTERVENTIONS:
Drug: sargramostim GZ402664 — Pharmaceutical form: lyophilized powder in vial
  Route of administration: subcutaneous
  Other Names: Leukine

SUMMARY:
Primary Objective:

Measure the proportion of patients who develop binding and neutralizing antibodies in the blood after treatment with sargramostim following induction/reinduction chemotherapy.

Secondary Objectives:

* Assess the time after treatment at which the antibodies develop and the level of antibodies is measured after the first dose.
* Measure the levels of immunoglobulin protein.
* Assess the impact of any immune response on safety and the duration of low white blood cell count.

DETAILED DESCRIPTION:
The total study duration for a participant is up to 6 months from 1st dose of sargramostim or until the antibodies level return to baseline or up to 24 months if antibodies test is positive at month 6.

ELIGIBILITY:
Inclusion criteria :

* Able to provide informed consent.
* Newly diagnosed acute myeloid leukemia (AML) to be treated with standard of care induction chemotherapy as per local policy.
* Patients 55 to 70 years of age (inclusive).
* Negative serum pregnancy test within 30 days prior to receiving the first dose of induction chemotherapy in female participants who are <2 years postmenopausal or who are of childbearing potential and have agreed to begin or continue using an adequate method of contraception.

Exclusion criteria:

* Prior treatment with sargramostim or any leukocyte growth factor (LGF) product.
* Prior myelodysplastic syndrome (MDS).
* Known central nervous system (CNS) leukemic involvement diagnosed by cytologic findings in cerebrospinal fluid and/or by computed tomography (CT) or magnetic resonance imaging (MRI).
* Out of range (>2x normal) laboratory values.
* Clinically important medical conditions unrelated to AML as determined by the Investigator.
* Eastern Cooperative Oncology Group (ECOG) performance status >2.
* Bone marrow blasts ≥5% on marrow examination following induction or reinduction chemotherapy.
* History of allergy to yeast products, recombinant human granulocyte/macrophage-colony-stimulating factor, or any component of sargramostim.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-02 (Estimated); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who develop antibodies (binding antibodies and neutralizing antibodies) | 1 month after 1st dose of sargramostim
Proportion of patients who develop antibodies (binding antibodies and neutralizing antibodies) | 2 months after 1st dose of sargramostim
Proportion of patients who develop antibodies (binding antibodies and neutralizing antibodies) | 3 months after 1st dose of sargramostim
Proportion of patients who develop antibodies (binding antibodies and neutralizing antibodies) | 6 months after 1st dose of sargramostim. If positive at month 6, this will be continued every 6 months until the values return to baseline or up to 24 months

SECONDARY OUTCOMES:
Assessment of antibodies (antibody detection and antibody titers) | 1 month after 1st dose of sargramostim
Assessment of antibodies (antibody detection and antibody titers) | 2 months after 1st dose of sargramostim
Assessment of antibodies (antibody detection and antibody titers) | 3 months after 1st dose of sargramostim
Assessment of antibodies (antibody detection and antibody titers) | 6 months after 1st dose of sargramostim. If positive at month 6, this will be continued every 6 months until the values return to baseline up to 24 months
Assessment of immunoglobulin levels | 1 month after 1st dose of sargramostim
Assessment of immunoglobulin levels | 2 months after 1st dose of sargramostim
Assessment of immunoglobulin levels | 3 months after 1st dose of sargramostim
Assessment of immunoglobulin levels | 6 months after 1st dose of sargramostim. If antibodies are positive at month 6, the level of immunoglubolins will be assesed every 6 months until the antibodies level return to baseline or up to 24 months
Proportion of patients with adverse events | Up to 24 months
Duration of neutropenia (time from initiation of sargramostim to recovery of ANC to ≥1500/mm^3) | Up to 42 days after first day of sargramostim administration

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi